CLINICAL TRIAL: NCT01225679
Title: Late-onset, Insidious Course and Invasive Treatment of Congenital Central Hypoventilation Syndrome in a Case With the Phox2B Mutation
Brief Title: Late-onset Congenital Central Hypoventilation Syndrome and the Mutation of Phox2B Gene
Acronym: CCHS
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, MD, PhD, Associação Fundo de Incentivo à Pesquisa
Other Study IDs: 512947
Record Dates: First submitted 2010-07-07; First posted 2010-10-21 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Congenital Central Hypoventilation Syndrome
Keywords: Congenital Central Hypoventilation Syndrome; Phox2B gene; invasive ventilation; genetics; late-onset; sleep; central sleep apnea
MeSH Terms: conditions — Congenital central hypoventilation syndrome; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Human
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- polysomnography: Overnight supervised polysomnography (Embla System®) was performed in a sleep laboratory, which included capnometry. Arterial blood gas analysis was performed by radial arterial puncture. Ventilatory response to progressive hypercapnia was measured using the Read breathing technique. Briefly, subjects rebreathed into an air tight 5-L bag containing a mixture of 8% carbon dioxide (CO2) and 40% oxygen (O2). The spirometer technology used to monitor ventilation was based on a bi-directional rotating vane principle (flow sensitive). A continuous record of CO2 concentration in the expired gas was obtained by a CO2 analyzer within the circuit. The ventilatory hypercapnic drive was calculated from the slope produced by changes in ventilation (L. min-1) and changes in end-tidal PCO2.
  Interventions: Device: positive airway pressure, Non-invasive mechanic ventilation

INTERVENTIONS:
Device: positive airway pressure, Non-invasive mechanic ventilation — Vpap: 16 cm H2O inspiratory and 8 cm H2O expiratory pressures, 20 irpm.
  Mechanic ventilation: tidal volume of 850 ml; 16 irpm; inspiratory pressure of 40 mmHg; PEEP: 5 cm H2O.
  Other Names: There is no other intervention description

SUMMARY:
Congenital central hypoventilation syndrome (CCHS) is a rare disorder of respiratory control characterized by ventilatory impairment that results in arterial hypoxemia. Although patients typically present this disease as newborns and rarely in later infancy, there have been reports of patients presenting with CCHS in adulthood.

The present study reports a unique familial case in which the father (proband) presented late-onset CCHS with an expansion mutation of the Phox2B gene that was confirmed by genetic analysis. Surprisingly, the proband did not report any manifestation of the disease during childhood, and the disease progressed following an insidious course until adulthood. At the time of diagnosis, he did not present signs of pulmonary hypertension and right-side heart failure. The patient responded well to nocturnal invasive ventilation. In contrast, his son presented CCHS as a newborn with the full complement of symptoms while his daughter did not.

The present report shows that CCHS cases characterized by a mutated Phox2 gene can progress without many symptoms and that the treatment approach used here was efficient for controlling the course of the disease. Furthermore, this case indicates that incomplete penetrance can occur. Genetic screening of family members is mandatory to evaluate the reproductive risk of the disease, especially because asymptomatic mutation carriers may be at high risk to develop the disease and transmit it to the next generation.

DETAILED DESCRIPTION:
Congenital central hypoventilation syndrome (CCHS) is a rare disorder of respiratory control characterized by ventilatory impairment that results in arterial hypoxemia. This condition worse during sleep and occurs in patients with normal mechanical properties of the lung. It is diagnosed in the absence of primary neuromuscular disease, identifiable brainstem lesions, and other sleep disturbances or substance use.

Amiel et al. (2003) identified a mutation in the Phox2B gene associated with CCHS, characterized by 5 to 9 alanine expansions within a 20-residue polyalanine region in exon 3 of the Phox2B gene. Several reports confirmed the findings of Amiel et al., supporting the view that this gene is a master switch for the development of the autonomic nervous system network linked to respiratory control. Transgenic animals carrying the human Phox2B mutation develop a similar phenotype and lack glutamatergic neurons located in the parafacial region in the brainstem, which are involved in breathing control.

Although patients typically present with CCHS as newborns and rarely in later infancy, there have been reports of patients presenting with CCHS in adulthood. In cases of late-onset CCHS, most patients report having had some symptoms since childhood, and they have parents with a history of CCHS. Symptoms of right-side heart failure are generally observed at the time of diagnosis, and nocturnal noninvasive ventilation is frequently indicated.

The present study reports a unique familial case of CCHS in which the father (proband) presented late-onset CCHS linked to a Phox2B gene expansion mutation. The presentation, course of development and treatment response for this patient was unique His son presented CCHS as a newborn, while his daughter did not.

ELIGIBILITY:
Inclusion Criteria:Family member

Exclusion Criteria:NA

Min Age: 5 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: familial case in which the father (proband) presented late-onset CCHS with an expansion mutation of the Phox2B gene that was confirmed by genetic analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Describe the clinical case apresentation | Years of evolution

CONTACTS AND LOCATIONS:
Overall Officials: Lia Rita A Bittencourt, PhD, Principal Investigator — Universidade Federal de São Paulo/UNIFESP
Locations (1):
- Disciplina de Medicina e Biologia do Sono, Departamento de Psicobiologia, Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil